CLINICAL TRIAL: NCT04262635
Title: A Phase III, Multicenter, Open-label, Randomized Study to Assess the Efficacy and Safety of Cetuximab Plus Capecitabine Versus Cetuximab as Maintenance Treatment Following First-line Induction Treatment With FOLFOX and Cetuximab in Chinese Patients With RAS and BRAF Wild-type Metastatic Colorectal Cancer
Brief Title: Cetuximab Plus Capecitabine as Maintenance Treatment in RAS and BRAF wt Metastatic Colorectal Cancer
Acronym: C-CLASSIC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Rui-hua Xu, MD, PhD, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-CLASSIC
Record Dates: First submitted 2020-02-05; First posted 2020-02-10 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ArmA Cetuximab plus Capecitabine (Experimental): Maintenance therapy with Cetuximab as intravenous (IV) infusion at the dose of 500 mg/m2, given every 2 weeks (Q2W); plus capecitabine in 2-week cycles until progressive disease, death from any cause, unacceptable toxicity or informed consent withdrawal
  Interventions: Drug: Cetuximab, Capecitabine
- ArmB Cetuximab (Active Comparator): Maintenance therapy with Cetuximab as intravenous (IV) infusion at the dose of 500 mg/m2, given every 2 weeks (Q2W) until progressive disease, death from any cause, unacceptable toxicity or informed consent withdrawal
  Interventions: Drug: Cetuximab

INTERVENTIONS:
Drug: Cetuximab, Capecitabine — Maintenance treatment ( ArmA )
  Arms: ArmA Cetuximab plus Capecitabine
Drug: Cetuximab — Maintenance treatment ( ArmB )
  Arms: ArmB Cetuximab

SUMMARY:
This is an open-label, multicenter, randomized study to be conducted in Chinese patients with RAS and BRAF wild-type mCRC. Patients who have already completed 9 cycles of standard first-line induction treatment, without discontinuation for toxicity, of cetuximab or fluorouracil or oxaliplatin,, and achieved disease control (including CR/PR and SD), and are progression free at the end of Cycle 9 will be assigned to 2 maintenance treatment groups by randomization in a 1:1 ratio to receive cetuximab + capecitabine (Arm A) or cetuximab alone (Arm B). The randomization will be stratified by induction treatment response (complete response [CR]+ partial response [PR] versus stable disease [SD]) and primary tumor location (left side only versus right side). All patients from Arm A and Arm B will be treated until progressive disease, death from any cause, unacceptable toxicity or informed consent withdrawal (whichever occurs earlier).

DETAILED DESCRIPTION:
Coz COVID-19 limited, C-CLASSIC was terminated recruitment on 31Dec2022. Total screen 100 subjects and enroll 80 subjects. All subjects in study will be treatment until meet study endpoint. Then study related subject follow up, data collect, clinical study report will be continued as planned.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent prior to performance of any study procedure.
2. Patient must be ≥18 years of age, at the time of signing the informed consent.
3. Patients who have histologically or cytologically confirmed adenocarcinoma of the colon or rectum, excluding appendix carcinoma or anal canal carcinoma, with RAS and BRAF wild-type mutation status.
4. Patients who received only FOLFOX plus cetuximab as first-line induction treatment after diagnosis of mCRC.
5. Having completed FOLFOX plus cetuximab for 9 cycles as induction treatment (in the first cycle, they could be treated with FOLFOX alone for waiting the results of genetic test) without discontinuation for toxicity, of cetuximab or fluorouracil or oxaliplatin and achieved disease control (including CR/PR and SD) and are progression free at the start of maintenance therapy.
6. At least one lesion(s), which is considered as unresectable at start of maintenance therapy (mCRC patients with resectable lesion(s) after induction treatment can be enrolled if they are willing to choose maintenance therapy). Patients who achieved CR and had no measurable lesion after induction treatment can be enrolled in this study.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
8. Life expectancy of at least 12 weeks in the opinion of the investigator.
9. Laboratory requirements

   * Neutrophils ≥1.5×109/L, platelets ≥75×109/L, and hemoglobin ≥9 g/dL;
   * Total bilirubin ≤1.5×upper limit of normal (ULN); aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT) and/or alanine aminotransferase (ALT)/serum glutamic-pyruvic transaminase (SGPT)

     * 2.5×ULN (≤5×ULN in case of liver metastases); alkaline phosphatase
     * 2.5×ULN (≤5×ULN in case of liver metastases, ≤10×ULN in case of bone metastases); lactate dehydrogenase (LDH) <1500 U/L;
   * Creatinine clearance (calculated according to Cockcroft and Gault) >60 mL/min or serum creatinine ≤1.5×ULN.

Exclusion Criteria:

1. Having received chemotherapy for mCRC other than induction therapy with FOLFOX plus cetuximab, except for adjuvant therapy that has ended >9 months (oxaliplatin- based chemotherapy) or >6 months (oxaliplatin-free chemotherapy), prior to the start of the induction treatment.
2. Other concurrently active malignancies, excluding malignancies that are disease free for more than 5 years or carcinoma-in-situ deemed cured by adequate treatment. Patients who are definitely detected as dMMR/MSI-H at the start of induction therapy.
3. Known brain metastasis or leptomeningeal metastasis. Patients with neurological symptoms should undergo brain computed tomography (CT)/ magnetic resonance imaging (MRI) to exclude metastases.
4. Unresolved toxicity greater than or equal to Common Terminology Criteria for Adverse Events (CTCAE) Grade 2 attributed to any prior therapies (excluding anemia, alopecia, skin pigmentation). Patients with platinum induced neurotoxicity greater than or equal to CTCAE Grade 3 should be excluded.
5. Ascites, pleural effusion or pericardial fluid requiring drainage in last 4 weeks.
6. Intestinal obstruction, major gastrointestinal hemorrhage or other diseases not suitable for maintenance treatment in this study as assessed by the investigator within 2 weeks prior to enrollment.
7. Diabetes and hypertension as assessed by the investigator as not eligible for the subsequent maintenance treatment in this study.
8. Myocardial infarction within the last 12 months, severe/unstable angina, symptoms of class III or IV congestive heart failure per New York Heart Association (NYHA) classification.
9. Previous hypersensitivity to any of the study drugs (cetuximab or capecitabine).
10. Deficiency in dihydropyrimidine dehydrogenase (DPD) as manifested by known medical history of fluorouracil adverse reactions.
11. Known infection with human immunodeficiency virus (HIV), acquired immunodeficiency syndrome (AIDS)-related illness, or active hepatitis B (positive HBsAg and HBV-DNA ≥ 2000 IU/mL or 104 copies/mL) or hepatitis C. Patients with previously confirmed COVID-19 infection, including severe, mild, asymptomatic, and recovered patients.
12. Patients with active autoimmune disorders requiring treatment or history of organ transplantation requiring immunosuppressive therapy.
13. Psychiatric disease that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results.
14. Treatment with any of the following within the specified time frame prior to study drug administration

    * Major surgery within 4 weeks (excluding diagnostic biopsy, the surgical incision should be fully healed prior to study drug administration);
    * Radiotherapy within 4 weeks;
    * Anti-cancer therapy other than protocol-specified induction therapy or participation in other clinical studies within 4 weeks.
    * Anti-tumor traditional Chinese medicine within 2 weeks (such as Cantharidin, Cinobufacini).
15. Pregnant (as determined by serum human chorionic gonadotropin [hCG] test) or lactating female, or female planning to become pregnant during treatment and for 2 months after the end of treatment with cetuximab and 6 months after the end of capecitabine. Woman of childbearing potential (WOCBP) with either positive or no pregnancy test at baseline. WOCBP or sexually active men not willing to use contraception during study and for at least 3 months after completion of cetuximab and 6 months after completion of capecitabine. Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential.
16. Presence of other serious disease or social circumstances that precludes patient enrollment in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-09-24 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy: Maintenance PFS | From Baseline to primary completion date, about 42 months
  mPFS from randomization to PD or death from any cause

SECONDARY OUTCOMES:
Number of Participants With Adverse Events During Treatment Period | From Baseline to primary completion date, about 42 months
  AEs included SAEs and non-serious AEs. Causality to study treatment was determined by the investigator. Severity was graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Number of Participants With Clinical Laboratory Abnormalities During Treatment Period | From Baseline to primary completion date, about 42 months
  Clinical laboratory tests include hematology, electrolyte and clinical chemistry.
Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-C30 (EORTC QLQ-C30) | From Baseline to primary completion date, about 42 months
  Quality of life is assessed using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) C30. It will be evaluated at Screening, Tumor Assessment Visit and End of Treatment visit.
Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-CR29 (EORTC QLQ-CR29) | From Baseline to primary completion date, about 42 months
  Quality of life in patients with colorectal cancer is assessed using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) CR29. It will be evaluated at Screening, Tumor Assessment Visit and End of Treatment visit.
Overall Survival | From Baseline to primary completion date, about 42 months
  Time from randomization to death from any cause

OTHER OUTCOMES:
Change from Baseline in Mutation Status of Selected Genes tested by Next-Generation Sequencing during Treatment Period | From Baseline to primary completion date, about 42 months
  Mutation status of selected genes (include but are not limited to KRAS, NRAS, BRAF, HER2, PI3K, NTRK, POLE, etc ) is assessed using Next-Generation Sequencing Method. It will be evaluated at Screening and End of Treatment visit with peripheral blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, MD, Study Chair — Sun Yat-sen University
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No